CLINICAL TRIAL: NCT05920135
Title: First-in-Human Study of BBT-207 in Advanced Non-Small Cell Lung Cancer Harboring EGFR Mutation After Treatment With EGFR TKI
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BBT207-ONC-001
Record Dates: First submitted 2023-05-26; First posted 2023-06-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-11

CONDITIONS: EGFR Mutant Advanced Non-Small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a; Dose escalation at various dose levels in patients with EGFR TKI sensitizing mutation (Experimental)
  Interventions: Drug: BBT-207
- Phase 1b; At 2 recommended dose levels of BBT-207 in patients with EGFR C797S mutation (Experimental)
  Interventions: Drug: BBT-207
- Phase 2; At the recommended phase 2 dose of BBT-207 in patients with EGFR C797S mutation (Experimental)
  Interventions: Drug: BBT-207

INTERVENTIONS:
Drug: BBT-207 — BBT-207 given orally alone

SUMMARY:
This is an open label, multi-center, Phase 1/2 study evaluating the safety, tolerability, PK, PD, and preliminary efficacy (antitumor activity) of BBT-207. It will consist of 3 parts; dose escalation, recommended phase 2 dose selection, and dose expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed Stage III (locally advanced) NSCLC not amenable to curative therapy or stage IV NSCLC.
2. Patients must have received treatment with at least 1 third-generation EGFR TKI (eg, Osimertinib, Lazertinib).
3. Confirmation that the tumor harbors an EGFR mutation as follows:

   1. Phase 1a (Dose Escalation): Confirmation that the tumor harbors an EGFR mutation known to be associated with EGFR TKI sensitivity (exon 19 deletion or L858R).
   2. Phase 1b (RP2D Selection): Have complex EGFR mutations containing C797S confirmed.
   3. Phase 2 (Dose Expansion): Have complex EGFR mutations containing C797S confirmed by a central laboratory.
4. Documented partial or complete response (CR) or durable (at least 16 weeks) stable disease, based on the RECIST criteria, after treatment of an EGFR TKI.
5. Radiological documentation of disease progression or intolerance to a previous continuous (at least 30 days) treatment with an approved EGFR TKI therapy (including, but not limited to osimertinib, afatinib, dacomitinib, gefitinib, or erlotinib).
6. All patients must have documented radiological progression or intolerance to the last treatment administered prior to enrolling in the study.
7. Has Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
8. Adequate organ function test result.
9. All standard therapeutic options have been exhausted, refused by the patient, or are contraindicated; or the patient is deemed by the investigator not to be an appropriate candidate for standard-of-care treatment (as defined in the country of participation).

Exclusion Criteria:

1. Has symptomatic brain or spinal cord metastases with exceptions.
2. Any of the following cardiac conditions within the last 6 months from the first dose of study treatment:

   1. Unexplained or cardiovascular cause of presyncope or syncope, tachycardia, ventricular fibrillation, or sudden cardiac arrest.
   2. Prolonged corrected QT interval (mean resting corrected QT interval using Fridericia's formula [QTcF] >470 msec from 3 ECGs).
   3. Clinically significant, uncontrolled, cardiovascular disease including congestive heart failure grade 3 or 4 according to the New York Heart Association classification; myocardial infarction or unstable angina, uncontrolled hypertension, or clinically significant, uncontrolled arrhythmias, including bradyarrhythmia that may cause QT prolongation (eg, Type II second degree heart block or third-degree heart block).

   <Prior or Concomitant Anticancer Therapy>
3. An EGFR TKI, including but not limited to osimertinib, afatinib, dacomitinib, gefitinib, or erlotinib within 8 days of the first dose of study treatment.
4. Small molecule targeted inhibitor other than EGFR inhibitor class or cytotoxic chemotherapy within 14 days, or biologic anticancer medicine (cytokines or antibodies, etc.) within 28 days (before the initiation of BBT-207 treatment) for the systemic treatment of advanced NSCLC.
5. Has toxicities from previous anticancer therapies that have not resolved to baseline levels or to CTCAE grade ≤1, with the exception of alopecia and peripheral neuropathy.
6. Has had radiotherapy within 14 days before the initiation of study treatment. Note: Palliative radiotherapy for pain can be administered at any time before the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
[Phase 1a dose escalation] Determine Recommended Dose Range | Approximately 12 months
  RDR determination: between the minimal reproducibly active dose and the maximum tolerated dose or maximum administered dose. Based on the totality of the data including toxicity/tolerability, efficacy, PK, and PD
[Phase 1a dose escalation] Incidence of Treatment-Emergent Adverse Events, Adverse Events of Special Interest, Serious Adverse Events, and ≥grade 3 laboratory abnormalities. | Throughout study completion, approximately 12 months
  Type, frequency, and severity of TEAEs according to NCI Common Terminology Criteria for Adverse Events Version 5.0 criteria.
[Phase 1b Recommended Phase 2 Dose selection] Determine the RP2D | Approximately 12 months
  RP2D determination: The Safety Monitoring Committee will determine the RP2D based on the totality of the data including overall safety, pharmacokinetic, pharmacodynamic, and preliminary antitumor activity including the percentage of patients with PR or CR based on RECIST Version 1.1.and duration of response.
[Phase 2 dose expansion] Evaluate preliminary antitumor activity | Approximately 12 months
  ORR defined as the percentage of patients with PR or CR based on RECIST Version 1.1.

SECONDARY OUTCOMES:
[Phase 1a, Phase 1b, Phase 2] observed maximum plasma concentration after administration [Cmax] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] time to reach the observed maximum (peak) concentration [Tmax] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] area under the plasma concentration-time curve from time zero to dosing interval [AUC0-τ] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] Area under the concentration-time curve from time zero to the time with last measurable concentration [AUC0-t] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] area under the concentration-time curve from time zero extrapolated to infinity [AUC0-∞] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] terminal elimination half-life [t½] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] terminal elimination rate constant [λz] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] apparent clearance following extravascular administration [CL/F] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] apparent volume of distribution following extravascular administration [Vz/F] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] accumulation ratio [Rac] for Cmax and area under the plasma concentration-time curve [AUC] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b, Phase 2] observed trough plasma concentration at the dosing interval [Ctrough] | Up to Cycle 2 Day 2 (each cycle is 21 days)
[Phase 1a, Phase 1b] ORR defined as the percentage of patients with PR or CR based on RECIST Version 1.1 | Approximately 12 months
[Phase 1a, Phase 1b, Phase 2] DCR per RECIST Version 1.1, measured as percentage of patients with CR + PR + (SD ≥16 weeks) | Approximately 12 months
[Phase 1a, Phase 1b, Phase 2] Time to Response [TTR] per RECIST Version 1.1 | Approximately 12 months
[Phase 1a, Phase 1b, Phase 2] Duration of Response [DOR] defined as the time from the first dose of BBT207 to disease progression or death in patients who achieve complete or partial response per RECIST Version 1.1 | Approximately 12 months
[Phase 1a, Phase 1b, Phase 2] Progression Free Survival [PFS] defined as the time from the first dose of BBT-207 until the date of first documented progressive disease or death due to any cause, whichever occurs first per RECIST Version 1.1 | Approximately 12 months
[Phase 2] Overall Survival [OS] defined as the time from the first dose of BBT-207 until the date of death due to any cause | Approximately 3 years
[Phase1b, Phase2] Incidence of Treatment-Emergent Adverse Events, Adverse Events of Special Interest, Serious Adverse Events, and ≥grade 3 laboratory abnormalities. | Throughout study completion, approximately 12 months
  Type, frequency, and severity of TEAEs according to NCI Common Terminology Criteria for Adverse Events Version 5.0 criteria.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul